CLINICAL TRIAL: NCT03280745
Title: Hypertonic Saline for Fluid Resuscitation After Cardiac Surgery
Acronym: HERACLES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201706011.1
Record Dates: First submitted 2017-08-23; First posted 2017-09-12 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases; Valvular Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Intervention Model Description: At admission to the ICU patients will receive 5ml/kg body weight of 7.3% NaCl or 0.9% NaCl by infusion pump over 60 minutes. If necessary, fluid resuscitation will be performed with Ringer's lactate to normalize peripheral perfusion and to allow weaning of vasopressors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7.3% NaCl (intervention) (Active Comparator): At admission to the ICU patients will receive 5ml/kg body weight of 7.3% NaCl NaCl by infusion pump over 60 minutes.
  Interventions: Drug: Hypertonic saline
- 0.9% NaCl (comparator) (Active Comparator): At admission to the ICU patients will receive 5ml/kg body weight of 0.9% NaCl by infusion pump over 60 minutes.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Hypertonic saline — At admission to the ICU patients will receive 5ml/kg body weight of 7.3% NaCl by infusion pump over 60 minutes.
  Other Names: 7.9% NaCl
  Arms: 7.3% NaCl (intervention)
Drug: 0.9% saline — At admission to the ICU patients will receive 5ml/kg body weight of 0.9% NaCl by infusion pump over 60 minutes.
  Other Names: normal saline
  Arms: 0.9% NaCl (comparator)

SUMMARY:
Background: Volume replacement strategies and type of fluid used in patients undergoing cardiac surgery have changed during the last years. Currently used crystalloid solutes have a variable composition and a major impact on organ function and outcome. Additionally critically ill patients are prone to fluid overload, which is despite common perception, not a benign occurrence as it is associated with prolonged ICU- and hospital length of stay and increased mortality rates. Fluid resuscitation using bolus or continuous infusion of hypertonic saline was used for more than thirty years. Only a few studies have been conducted so far, but they showed that infusion of hypertonic saline results in less volume administered, increased renal function less weight gain in critically ill patients when compared to other crystalloids.

Aim: This preliminary randomized controlled double-blind study aims to identify whether fluid resuscitation using hypertonic saline (HS) when used in addition to lactated Ringers solution results in less total fluid amount administered in patients following cardiac surgery. Additionally we want to evaluate whether the use of hypertonic saline results less need for pharmacological cardiocirculatory support, increased renal function, less postoperative volume overload shortened post-cardiac bypass immune suppression and increased postoperative outcomes.

Study intervention: At admission to the ICU patients will receive 5ml/kg body weight of 7.3% NaCl or 0.9% NaCl by infusion pump over 60 minutes. If necessary, fluid resuscitation will thereafter be performed with Ringer's lactate to normalize peripheral perfusion and to allow weaning of vasopressors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery for ischemic or valvular heart disease

Exclusion Criteria:

* Patients unable to give informed consent
* Patients with age <18 years
* Pregnancy or breastfeeding
* Left-ventricular ejection fraction (LVEF) < 30% preoperatively
* Preexisting renal insufficiency with an eGFR <30 ml/min/1.73m2
* Patients with postoperative circulatory support devices such as LVAD, IABP, Impella, ECMO
* Preexisting serum sodium of >145mmol/l or <135 mmol/L
* Preexisting serum chloremia >107mmol/l or < 98 mmol/L
* Systemic steroid therapy (at any dose at time of inclusion)
* Chronic liver disease (bilirubin >3 mg.dl)
* Any signs of infection or sepsis defined as clear clinical evidence for active infection or current antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
total cumulative amount of fluids infused | daily until ICU discharge, max until postoperative day 90

SECONDARY OUTCOMES:
postoperative weight gain | until postoperative day 6
total postoperative cumulative urinary output | daily until ICU discharge, max until postoperative day 90
total cumulative dose of inopressors per kg bodyweight /hour | until ICU discharge, max until postoperative day 90
  cumulation of norepinephrine and epinephrine
time on inopressors | from ICU admission until stop of inopressors, max until postoperative day 90
  norepinephrine and/or epinephrine
variation in renal function markers | until postoperative day 6
  renal damage maker (TIMP2-IGFB, creatinine)
variation in acid-base homeostasis | until postoperative day 6
  pH, base excess, lactate, bicarbonate, electrolytes
variation in immune function | until postoperative day 6
  mHLA-DR
time on the ventilator | from ICU admission until time of extubation, maximum 90 days
occurence of infection | occurence of infection during the index hospitalisation or subsequent admissions due to infection upto 90 postoperative days
length of stay | time to ICU/hospital-discharge however long this may take, maximum 90 days
  time to ICU/hospital-discharge
readmissions to the ICU | readmissions to the ICU within postoperative 90 days
mortality | until postoperative day 90

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Schefold, MD, Study Director — Department of Intensive Care, Inselspital, Bern University Hospital, Bern, Switzerland
Locations (1):
- Department of Intensive Care, Bern University Hospital and University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfortmueller CA, Messmer AS, Hess B, Reineke D, Jakob L, Wenger S, Waskowski J, Zuercher P, Stoehr F, Erdoes G, Luedi MM, Jakob SM, Englberger L, Schefold JC. Hypertonic saline for fluid resuscitation after cardiac surgery (HERACLES): study protocol for a preliminary randomised controlled clinical trial. Trials. 2019 Jun 14;20(1):357. doi: 10.1186/s13063-019-3420-6. PMID 31200756